CLINICAL TRIAL: NCT02009020
Title: Evaluation of a Non-invasive Device to Measure Blood Pressure and Difference in Pulse Pressure (dPP) Intraoperatively
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Verena Schnupp, M.D., Johannes Gutenberg University Mainz
Other Study IDs: 837.531.11 (8073)
Record Dates: First submitted 2013-12-04; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Blood Pressure

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Dynamic parameters like pulse pressure Variation (PPV) , synonymous: difference in pulse pressure (dPP), can predict fluid responsiveness reliably (Marik PE et al, Crit Care Med 2009; 37:2642-7). An arterial line is required for assessment of dPP. On a modified Penaz technique, a non-invasive measurement device is now available commercially. In this study, the reference technique based on arterial measurement and a respiratory variation monitor (Pestel G et al, Anesth Analg 2009; 108:1823-9) was compared to the non-invasive device a clinical setting. At defined time points, systolic, diastolic, mean arterial blood pressure and dPP were compared using Bland-Altmann Analysis (Bland JM, Altman DG, Lancet 1986; 1: 307-10)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 80 years old
* Written informed consent obtained
* Patients scheduled for elective urological or abdominal surgery procedures in supine position
* qualifying for arterial line

Exclusion Criteria:

* pregnancy
* cardiac insufficiency (NYHA 4, EF < 25 %)
* coronary artery disease (CCS 4)
* coagulopathy
* symptoms of infection or sepsis
* malignant hyperthermia
* absence of sinus rhythm
* BMI > 30
* M. Raynaud

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective abdominal or urological surgery
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Comparison between arterial line and non-invasive device for blood pressure and difference in pulse pressure measurement | intraoperatively
  Systolic, diastolic, mean blood pressure and difference in pulse pressure are measured intraoperatively with a non-invasive device and the reference technique. The values are compared using Bland-Altmann Analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaetsmedizin - Johannes Gutenberg University Mainz (Department of Anesthesiology), Mainz, Germany

REFERENCES:
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Pestel G, Fukui K, Hartwich V, Schumacher PM, Vogt A, Hiltebrand LB, Kurz A, Fujita Y, Inderbitzin D, Leibundgut D. Automatic algorithm for monitoring systolic pressure variation and difference in pulse pressure. Anesth Analg. 2009 Jun;108(6):1823-9. doi: 10.1213/ane.0b013e3181a2a8bf. PMID 19448207
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172